CLINICAL TRIAL: NCT05753345
Title: Aquatic Therapy for Children With Neuromotor Deficits
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Collaborators: Franklin County Board of Developmental Disabilities (Unknown)
Responsible Party: Principal Investigator, Erika Kemp, Assistant Professor, Clinical, Ohio State University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022H0340
Record Dates: First submitted 2023-02-03; First posted 2023-03-03 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-12

CONDITIONS: Cerebral Palsy; Hypoxia, Brain
MeSH Terms: conditions — Cerebral Palsy; Hypoxia, Brain | interventions — Aquatic Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention: aquatic occupational therapy (AquOTic-NM) (Experimental): aquatic occupational therapy 30 minutes, self care training 15 minutes
  Interventions: Behavioral: Aquatic therapy

INTERVENTIONS:
Behavioral: Aquatic therapy — Children receive aquatic occupational therapy twice a week for 10 weeks. 30 minutes of aquatic therapy in a warm water pool to increase upper extremity function and swim skills; 15 minutes of self care training to increase independence with dressing and showering.

SUMMARY:
The purpose of this study is to explore the feasibility, fidelity and acceptability of an aquatic therapy assessment and intervention for children ages 3-9 with neuromotor deficits such as cerebral palsy. The intervention takes place in a warm water therapy pool, twice a week for ten weeks and targets swim safety skills, upper extremity function and self care participation and performance.

DETAILED DESCRIPTION:
The purpose of this study is to explore the feasibility, fidelity and acceptability of an aquatic therapy assessment and intervention. The intervention will target swim safety skills, upper extremity function and self care participation and performance in children with neuromotor conditions such as cerebral palsy. The study includes an intake evaluation session, twenty sessions of aquatic therapy (twice a week for 10 weeks) and a post evaluation session. This takes place in Columbus, Ohio.

Each session will be a combination of land-based self care training and water-based upper extremity exercise and swim skill training. The intervention structure will include the following:

1. Self Care Session: Doffing clothing, preparing for swimming
2. Motor learning aquatic activities guided by individualized goals
3. Self Care session: Towel dry, rinse off, dressing

Individualized activities will be planned according to the individualized goals written for each child participant.

ELIGIBILITY:
Inclusion Criteria:

* 3-9 years for the children, 18+ for the parents/guardians.
* child with neuro-motor diagnosis (CP, hypoxia, etc.)
* child impairments in upper extremity function
* child deficits in performance of self care activities

Exclusion Criteria:

* compromised airway
* uncontrolled seizures

Ages: 3 Years to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 36 (Estimated)
Dates: Start 2023-01-09 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Change in Water Orientation Test Alyn (WOTA) | Baseline, immediately after the intervention
  performance based swim skill assessment
Change in Pediatric Evaluation of Disability Index, Computer Adaptive Text (PEDI-CAT) | baseline, immediately after the intervention
  parent reported questionnaire regarding child's self care skills
Change in Quality of Upper Extremity Skills Test (QUEST) | baseline, immediately after intervention
  performance-based assessment of upper extremity skills

SECONDARY OUTCOMES:
Change in Participation and Environment Measure (PEM-CY) | baseline, immediately after the intervention
  parent reported questionnaire of participation in home, school and community
Change in Canadian Occupational Performance Measure (COPM) | baseline, immediately after the intervention
  Parent perception of goals attained

CONTACTS AND LOCATIONS:
Locations (1):
- Erika Kemp, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No
Deidentified data maybe shared with researchers